CLINICAL TRIAL: NCT03782038
Title: A Prospective, Multi-center, Pilot Study to Evaluate the Safety and Efficacy of the Cytrellis Micro-Coring Device for the Treatment of Scars
Brief Title: Study to Evaluate the Efficacy of a Micro Coring Device for the Treatment of Scars of the Cytrellis Micro-Coring Device for the Treatment of Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cytrellis Biosystems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIS 700-00053
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Scars
Keywords: Acne Scars; Stretchmarks; Surgical Scars
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Micro-coring of scars with MCD (Experimental): Micro coring of acne scars and straie will be conducted in up to 3 treatments and followed 6 months post last treatment with MCD.
  Interventions: Device: MCD

INTERVENTIONS:
Device: MCD — Micro coring skin removal with automated coring device

SUMMARY:
A study to evaluate the safety and effectiveness of a micro coring device for the treatment of scars.

DETAILED DESCRIPTION:
The study subject population will consist to up to 30 subjects who meet the inclusion/exclusion criteria. All subjects will be monitored for a period of 6 months post last treatment.

An study results will be assessed on the following:

* POSAS - Patient Observer Scar Assessment
* ASAS - Acne Scar Severity Scale
* Subject Satisfaction Scale

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Fitzpatrick scale I-VI.
* Any type of scar except for keloid scars
* Able to provide written informed consent, understand and willing to comply with study related procedures and follow-ups.

Exclusion Criteria:

* Previous treatment of the scar tissue within last 6 months.
* Silicone, fat, collagen or synthetic material in the treatment area.
* History of keloid formation.
* Active smokers (smoking more than ½ pack per day) or having quit smoking (½ pack per day) for less than 3 months.
* Active, chronic, or recurrent infection.
* Compromised immune system (e.g. diabetes).
* Hypersensitivity to analgesic agents.
* Co-morbid condition that could limit ability to participate in the study or to comply with follow-up requirements.
* Pregnant or breastfeeding.
* Any issue that, at the discretion of the investigator, would contra-indicate the subject's participation.
* Any medication that may cause bleeding such as anticoagulants.
* Allergy to lidocaine and/or epinephrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-09-17 (Estimated); Study Completion 2019-11-21 (Estimated)

PRIMARY OUTCOMES:
Assess level of aesthetic improvement using POSAS scale 6 months post last treatment | 6 months post last treatment
  Assessing the improvement in the aesthetic appearance of the subject based on the POSAS scale comparing baseline to 6 months post last treatment. Parameters of vascularity, pigmentation, thickness, relief, and pliability, range from 1 to 10. normal skin =1; worst scar imaginable =10.
Assess level of aesthetic improvement using ASAS scale 6 months post last treatment | 6 months post last treatment
  Assessing the improvement in the aesthetic appearance of the subject based on the Acne Scar scale comparing baseline to 6 months post last treatment. Grades range 0-4. Clear =0; Very Mild=1; Mild= 2; Moderate= 3; Severe= 4

SECONDARY OUTCOMES:
Assess safety profile by recording all adverse events reported during study | 6 months post last treatment
  Adverse events will be recorded throughout the study

CONTACTS AND LOCATIONS:
Locations (1):
- Miami Dermatology & Laser Institute, Miami, Florida, United States